CLINICAL TRIAL: NCT01515930
Title: Computer-Delivered Motivational Intervention to Improve Teen Diabetes Management
Brief Title: Computerized Intervention of Parental Involvement in Diabetes Care of Their Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3M's Diabetes Study; R21DK089238 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Diabetes
Keywords: Parenting; Parental Monitoring; Diabetes; Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Caregiver and Active Child (Active Comparator): Parent & Child Computer-Delivered Motivational Intervention will be delivered to participants. A brief computer delivered behavior change counseling intervention for parents of children with diabetes to improve monitoring of diabetes care and a brief computer delivered behavior change counseling intervention for children with diabetes to improve completion of daily diabetes care.
  Interventions: Behavioral: Parent & Child Computer-Delivered Motivational Intervention
- Active Caregiver and Child Education (Experimental): Parent Computer-Delivered Motivational Intervention will be delivered to the parents only. A brief computer delivered behavior change counseling intervention for parents of children with diabetes to improve monitoring of diabetes care and a brief computer delivered informational session about diabetes related topics for their child with diabetes.
  Interventions: Behavioral: Parent Computer-Delivered Motivational Intervention
- Education Caregiver/Education Child (Active Comparator): Participants will receive computer-delivered information. A brief computer delivered information session about diabetes related topics for both the caregiver and the child with diabetes.
  Interventions: Behavioral: Computer-Delivered Information

INTERVENTIONS:
Behavioral: Parent Computer-Delivered Motivational Intervention — Motivational Interviewing (MI) is a client-centered, directive method for enhancing intrinsic motivation to change by exploring & resolving ambivalence, with a strong evidence for improving adolescent & adult health behaviors. Three motivational sessions will be provided by an animated character who delivers the intervention with high fidelity to MI principles. Small amounts of psychoeducation about potential improvements illness management that can result from parental monitoring of diabetes care will be integrated with more purely motivational elements. Mailings will be sent to participants to remind them of the reasons they gave as motivation & goals they set regarding monitoring diabetes care.
  Arms: Active Caregiver and Child Education
Behavioral: Parent & Child Computer-Delivered Motivational Intervention — Motivational Interviewing (MI) is a client-centered, directive method for enhancing intrinsic motivation to change by exploring & resolving ambivalence, with a strong evidence for improving adolescent & adult health behaviors. Three motivational sessions will be provided by an animated character who delivers the intervention with high fidelity to MI principles. Small amounts of psychoeducation about potential improvements illness management that can result from monitoring/completing diabetes care will be integrated with more purely motivational elements. Mailings will be sent to participants to remind them of the reasons they gave as motivation & goals they set regarding diabetes care.
  Arms: Active Caregiver and Active Child
Behavioral: Computer-Delivered Information — Computer-Delivered Information about issues related to living with diabetes that do not directly impact completing diabetes care.
  Arms: Education Caregiver/Education Child

SUMMARY:
The purpose of this study is to develop an intervention to increase parental motivation for supervision and monitoring youth diabetes care behavior. The intervention will be tested in three brief session in conjunction with regularly scheduled diabetes clinic visits and delivered through a computer program based in the principles of Motivational Interviewing.

DETAILED DESCRIPTION:
The study includes a development phase (Phase 1: development of the intervention followed by feasibility testing with 10 youth and 10 parents) and a pilot validation phase [Phase 2: pilot randomized clinical trial (RCT)] using a sample of 90 African American youth transitioning to independent diabetes care and their parents. In this phase, families will be randomly assigned to one of three study arms: parent motivation for monitoring and youth motivation for diabetes care (arm 1), parent motivation for monitoring and youth information (arm 2) or parent and youth information (arm 3). In phase 1 (development), youth and their caregivers will complete a one-time research visit where they use the program and provide feedback via a semi-structured interview regarding the usefulness of the content, its user-friendliness and make suggestions for changes to enhance acceptability. In phase 2 ( RCT), families will complete three intervention plus data collection visits and one additional data collection only visit. Research visits will be scheduled to coincide with appointments in the diabetes clinic to maximize convenience for families.

ELIGIBILITY:
Inclusion Criteria:

* African American race/ethnicity
* Age: 10 years 0 months - 12 years, 11 months
* Type 1 diabetes mellitus
* Diagnosed at least 6 months
* Patient of Children's Hospital of Michigan Diabetes Clinics
* English fluency, both verbal and written

Exclusion Criteria:

* Psychiatry/psychological diagnoses including cognitive impairment that would prevent the participant from understanding the data collection measures, (i.e. moderate or severe mental retardation) or the following psychiatric diagnoses: autism and schizophrenia. Youth with current suicidal intent are not enrolled until psychiatrically stable.
* Medical diagnoses that would result in atypical diabetes management i.e. cystic fibrosis. Other medical conditions that would not affect diabetes management, such as asthma, do not exclude the participant from study participation.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03-03 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
Diabetes Management Scale | Each of 3 intervention session, 3-4 month apart
  The Diabetes Management Scale (DMS) (Frey, Ellis, Naar-King et al., 2004) is a self-report questionnaire used to measure a broad range of diabetes management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision.

SECONDARY OUTCOMES:
Treatment Regulation Questionnaire | Each of 3 intervention session, 3-4 month apart
  Parental motivation to monitor the youth is measured by the Treatment Self-Regulation Questionnaire (TSRQ; Ryan & Connell (1989). The TSRQ evaluates why people engage in a health-relevant behavior and assesses the degree to which one's motivation for a particular behavior or set of behaviors is relatively autonomous or self-determined as compared to derived from external pressures or constraints.
Readiness Ruler | Each of 3 intervention session, 3-4 month apart
  Parent motivation to monitor the youth is also measured by the Readiness Ruler (Stott, Rollnick, & Pill, 1995). Since readiness to change behaviors is behavior specific, the items will be tailored to assess the behaviors most critical to parental monitoring of diabetes management. The response format is a visual analog scale (VAS) 10 mm in length. Written cues anchor the ends and middle of the scale. Respondents mark their "readiness" on the scale and the position on the line is measured in millimeters.
HbA1C Blood Test | Each of 3 intervention session, 3-4 month apart
  Metabolic control will be measured via hemoglobin A1c (HbA1c). HbA1c is an indirect and retrospective measure of average blood glucose levels over the previous two to three month period.
Parental Monitoring of Diabetes Care | Each of 3 intervention session, 3-4 month apart
  The Parental Monitoring of Diabetes Care scale (PMDC) is an 18 item, investigator-developed questionnaire that measures the frequency of parental monitoring and direct supervision of diabetes care tasks such as insulin administration, blood glucose testing, and dietary management.
Twenty-four Hour Recall Interview | Each of 3 intervention session, 3-4 month apart
  The Twenty-four Hour Recall Interview, developed by Johnson and colleagues (Freund, Johnson, Silverstein et al., 1991), has been used extensively in pediatric diabetes research for the assessment of illness management.
Blood Glucose Testing Frequency | Each of 3 intervention session, 3-4 month apart
  Objective data on mean daily frequency of blood glucose testing during the 14-day period prior to data collection will be obtained directly from blood glucose meters.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Ellis, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Idalski Carcone A, Ellis DA, Naar S, Ondersma SJ, Moltz K, Dekelbab B, Joseph CL. Enhancing parental motivation to monitor african american adolescents' diabetes care: development and Beta test of a brief computer-delivered intervention. JMIR Res Protoc. 2014 Sep 18;3(3):e43. doi: 10.2196/resprot.3220. PMID 25236503